CLINICAL TRIAL: NCT03454724
Title: A Multi Center Randomized Control Study of MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System in Treatment of Coronary Artery Disease Patients: MeRes - China.
Brief Title: Study of MeRes100 in the Treatment of Patient With Coronary Artery Disease.
Acronym: MeReS100-China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeRes-201706
Record Dates: First submitted 2018-01-15; First posted 2018-03-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: BioResorbable Vascular Scaffold System
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization of Study Device and Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MeRes100 BRS (Experimental): MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System indicated for the treatment of coronary artery disease along with standard percutaneous angioplasty procedure.
  Interventions: Device: MeRes100 Sirolimus-Eluting BioResorbable Vascular Scaffold System; Device: Xience EES Everolimus Eluting Coronary Stent System
- Xience EES (Active Comparator): Xience EES is a Everolimus Eluting Coronary Stent System indicated for the treatment of coronary artery disease along with standard percutaneous angioplasty procedure.
  Interventions: Device: MeRes100 Sirolimus-Eluting BioResorbable Vascular Scaffold System; Device: Xience EES Everolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: MeRes100 Sirolimus-Eluting BioResorbable Vascular Scaffold System — MeRes100 Sirolimus-Eluting BioResorbable Vascular Scaffold System used in the treatment of patients with coronary artery disease along with standard percutaneous angioplasty procedure.
Device: Xience EES Everolimus Eluting Coronary Stent System — Xience EES Everolimus Eluting Coronary Stent System indicated for the treatment of coronary artery disease along with standard percutaneous angioplasty procedure.

SUMMARY:
This is a Multi Center Randomized Control Study of MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System in treatment of approximately 484 subjects with Coronary Artery Disease in China. Eligible subjects shall have up to two de novo lesions in different epicardial vessels (One lesion in each coronary artery or it's major branch),Target lesion shall have visually estimated diameter stenosis ≥ 70% (or ≥ 50% and has clinical evidence of myocardial ischemia), lesion length ≤ 24mm, reference vascular diameter visually ≥ 2.75mm and ≤ 4.0mm. And subjects must meet all the study inclusion / exclusion criteria before enrolment in the study.All subjects shall accept clinical follow up at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post procedure.

DETAILED DESCRIPTION:
This is a Multi Center Randomized (MeRes:XIENCE=1:1) Control Study of MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System in treatment of approximately 484 subjects with Coronary Artery Disease in China. The post marketed XIENCE Everolimus Eluting Coronary Stent System will serve as the control device, to evaluate the safety and efficacy of MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System in coronary artery disease, and to support the product registration approval of the China Food and Drug Administration (CFDA).

Eligible subjects shall have up to two de novo lesions in different epicardial vessels ( One lesion in each coronary artery or it's major branch),Target lesion shall have visually estimated diameter stenosis ≥ 70% (or ≥ 50% and has clinical evidence of myocardial ischemia), lesion length ≤ 24mm, reference vascular diameter visually ≥ 2.75mm and ≤ 4.0mm. And subjects must meet all the study inclusion / exclusion criteria before enrolment in the study.

All the subjects shall accept angiography follow up at 12 months post procedure.

OCT subgroup ((N=80, 40 from test group and 40 from control group) shall accept follow up of OCT at immediately and 12 months post procedure. In segment late lumen loss at 12 months post procedure is the primary endpoint, and the percentage of stent strut neointimal coverage assessed with OCT at 12 months post procedure is the key secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Age ≥ 18 and ≤75years old, man or non-pregnant or non-lactating woman.
  2. Subjects with asymptomatic ischemic evidence, stable or unstable angina, or old myocardial infarction >7 days, suitable for selective PCI. Subjects without contraindications of coronary artery bypass grafting.
  3. Subjects be able to understand the purpose of this study, volunteer to participate and sign informed consent, willing to accept invasive imaging follow-up.

Angiographic inclusion criteria:

1. One de novo target lesion or up-to two de novo target lesions in different epicardial vessels: Different epicardial vessels are defined as left anterior descending artery (LAD) and its branches, left circumflex artery (LCX) arteries and its branches, and right coronary arteries (RCA) and its branches. Thus, for example, the subject must not have two target lesions required to be treated at the LAD and its branches at the same time.
2. Target lesion diameter stenosis ≥ 70% (or ≥ 50% simultaneously shall have clinical evidence of myocardial ischemia), and TIMI flow grade ≥1.
3. Target lesion length ≤ 24mm (estimated visually); reference vessel diameter between ≥ 2.75 mm to ≤ 4.00 mm.
4. Each target lesion can be fully covered by one scaffold.

Exclusion Criteria:

* General exclusion criteria:

  1. Any non-target lesion in coronary artery needs to be treated simultaneously or selectively (anticipation within 1 year), non-target lesion defined as any lesion that does not fulfill the inclusion/exclusion criteria.
  2. Any newly onset acute myocardial infarction within 1 week (< 7days) or, myocardial enzyme has not return to normal level (clinically non-significant) after myocardial infarction.
  3. Subject has undergone prior PCI within the target vessel during the last 12months or plans to receive another PCI within 6months or subject with history of CABG.
  4. Subjects with severe heart failure, such as ≥ grade III NYHA or left ventricular ejection fraction <30% (accessed by ECHO/ultrasound or left ventricular angiography).
  5. Blood tests shows the platelet count is less than 100 × 109 / L, or more than 700 ×109 / L, the white blood cells count is less than 3 × 109 / L.
  6. Pre-procedure severe liver or kidney functional damaged: serum creatinine> 1.5mg

     / dl (132.6μmol / L) or subject is receiving hemodialysis, ALT or AST were three times greater than the upper limit of normal.
  7. Subjects with bleeding tendency, active gastrointestinal ulcers, history of cerebral hemorrhage or history of subarachnoid hemorrhage, history within six months of ischemic stroke, contraindications of anti-platelet agents and anticoagulants treatment, and subjects cannot receive anti-thrombolytic therapy.
  8. Hypersensitive or allergic to antiplatelet drugs(such as aspirin and clopidogrel), anticoagulant drugs(such as heparin), contrast media, and scaffold components(such as PLLA，PDLLA, sirolimus, everolimus, iridium and platinum).
  9. The subject's life expectancy is less than 12 months.
  10. Subjects who anticipated in other drug or medical device clinical trial but haven't finished the primary endpoint evaluation visit.
  11. The investigators judged that subjects were poorly compliance and unable to complete the study as required.
  12. Subjects have accepted substantial organ transplant or ready to undergo organ transplant.
  13. Subjects have unstable arrhythmia, such as high-risk ventricular premature beats, and ventricular tachycardia.
  14. Subjects are receiving or planning to receive chemotherapy.
  15. Subjects have received or planning to receive radiotherapy.
  16. Subjects with immunosuppressive or autoimmune diseases, are receiving or planning to receive immunosuppressive therapy.
  17. Patients suffering from HIV, HBV or HCV infections
  18. Subjects are planning to receive or are receiving long-term anticoagulation therapy, such as heparin, warfarin and similar agents.
  19. Subjects are planning to accept selective surgery within 12 months, need to discontinue aspirin or clopidogrel (DAPT therapy).
  20. Subjects with diffuse peripheral vascular disease, cannot use 6F catheter.

Angiographic exclusion criteria:

1. Subjects with coronary artery triple vessel lesion in LAD, LCX or RCA, all need to be treated.
2. Target lesion locates in left main.
3. Target lesion locates in the aorto-ostial of RCA (within 3 mm of the origin of the RCA).
4. Target lesion locates within 3 mm of the origin of the LM, LAD and LCX.
5. Target lesion involving a bifurcation with a:

   1. Side branch ≥2.0 mm in diameter, or
   2. Side branch with diameter stenosis ≥ 50%, or
   3. Side branch requiring protection guide wire, or
   4. Side branch requiring pre-dilatation.
6. Anatomy proximal to or within the lesion that may impair delivery of the

   MeRes100TM or Xience EES, including:
   1. Extreme angulation (≥ 90°) proximal to or within the target lesion
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion
   3. Moderate or heavy calcification proximal to or within the target lesion
7. Target lesion involves a myocardial bridge.
8. Target vessel contains thrombus as indicated in the angiographic images or IVUS.
9. Target vessel has been previously treated with a stent at any time prior to the index procedure such that the MeRes100TM or XIENCE stent would need to cross the stent to reach the target lesion..
10. Target vessel has been previously treated with a stent and the target lesion is within 5 mm proximal to a previously treated lesion.
11. Chronic complete occlusive lesion (preoperative TIMI grade 0 flow).
12. Target lesion which prevents complete balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

    1. Residual %DS is < 40% (per visual estimation), ( ≤ 20% is strongly recommended).
    2. TIMI Grade-3 flow (per visual estimation).
    3. No angiographic complications (e.g., no-reflow, distal embolization, side branch closure).
    4. No dissections NHLBI grade D-F.
    5. No chest pain lasting > 5 minutes.
    6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
In-segment Late Lumen Loss | 12 Months
  Angiographic analysis for measuring Late Lumen Loss in both the treatment group

SECONDARY OUTCOMES:
The percentage of stent strut neointimal coverage assessed with OCT | 12 Months
  OCT analysis will be done to identify percentage of Neointimal coverage

CONTACTS AND LOCATIONS:
Overall Officials: Gao Runlin, MD, Principal Investigator — Fuwai Hospital CAMS

IPD SHARING:
Plan to Share IPD: No